CLINICAL TRIAL: NCT06579365
Title: Argentinean Registry on the Management of Helicobacter Pylori Infection
Acronym: ArgReg-Hp
Status: Recruiting | Type: Observational
Sponsor: University of Buenos Aires (Other)
Responsible Party: Principal Investigator, Oscar Laudanno, Chief Gastroenterology Department. Institute of Medical Research A Lanari, University of Buenos Aires. Faculty of Medicine, University of Buenos Aires
Other Study IDs: Registro Argentino H pylori
Record Dates: First submitted 2024-08-22; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: H.Pylori Gastrointestinal Disease; H Pylori Infection
Keywords: H pylori

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Helicobacter pylori (H pylori) is the main cause of chronic gastritis and peptic ulcer disease. In addition, is the main risk factor for gastric adenocarcinoma and mucosa-associated lymphoid tissue lymphoma. It is estimated that around 50% of the Argentinean population is infected with H pylori. The optimal management of H pylori remains unclear. In Argentina, most treatments are prescribed on an empiric basis, unaware of the bacterial antibiotic resistance profile.

Meta-analysis showed that susceptibility-guided treatment is not better than empirical treatment in first and second line treatment therapy if the most effective local regimens are prescribed. Updated information concerning local data is needed to design the best strategy to treat H pylori infection in order to reach high eradication rates and to introduce the principles of antimicrobial stewardship to reduce inappropriate antibiotic use.

The Argentinean Registry on H pylori (ArgReg-Hp) management was launched in May 2021 in order to obtain a large and representative sample of routine clinical practice of Argentinean gastroenterologist. Its main focus was to identify therapies that are highly effective and can be used empirically. Test of cure data is a surrogate method for susceptibility testing and resistance Primary aim To obtain a database registering systematically of a large and representative sample of routine clinical practice of Argentinean gastroenterologists in order to produce descriptive studies of the management of H. pylori infection.

Secondary aims To perform studies focused on epidemiology, efficacy and safety of the commonly used treatments to eradicate H. pylori.

The Argentinean Registry on H pylori management is a National , multicenter, prospective, non interventional registry recording data on H pylori management since May 2021. The ArgReg-Hp is promoted by Instituto de Investigaciones Médicas Alfredo Lanari (IDIM), Universidad de Buenos Aires and Club Argentino Estómago y duodeno (CADED).

Ethics: ArgReg-Hp was approved by the Ethics Committee IDIM, University of Buenos Aires as the reference IRB, and was approved by each center participant

DETAILED DESCRIPTION:
Helicobacter pylori (H pylori) is the main cause of chronic gastritis and peptic ulcer disease. In addition, is the main risk factor for gastric adenocarcinoma and mucosa-associated lymphoid tissue lymphoma. It is estimated that around 50% of the Argentinean population is infected with H pylori. The optimal management of H pylori remains unclear. Most treatments are prescribed on an empiric basis, unaware of the bacterial antibiotic resistance profile.

Meta-analysis showed that susceptibility-guided treatment is not better than empirical treatment in first and second line treatment therapy if the most effective local regimens are prescribed. Updated information concerning local data is needed to design the best strategy to treat H pylori infection in order to reach high eradication rates and to introduce the principles of antimicrobial stewardship to reduce inappropriate antibiotic use.

The Argentinean Registry on H pylori (ArgReg-Hp) management was launched in May 2021 in order to obtain a large and representative sample of routine clinical practice of Argentinean gastroenterologist. Its main focus was to identify therapies that are highly effective and can be used empirically. Test of cure data is a surrogate method for susceptibility testing and resistance Primary aim To obtain a database registering systematically of a large and representative sample of routine clinical practice of Argentinean gastroenterologists in order to produce descriptive studies of the management of H. pylori infection.

Secondary aims To perform studies focused on epidemiology, efficacy and safety of the commonly used treatments to eradicate H. pylori.

The Argentinean Registry on H pylori management is a National , multicenter, prospective, non interventional registry recording data on H pylori management since May 2021. The ArgReg-Hp is promoted by Instituto de Investigaciones Médicas Alfredo Lanari (IDIM), Universidad de Buenos Aires and Club Argentino Estómago y duodeno (CADED).

Ethics: ArgReg-Hp was approved by the Ethics Committee IDIM, University of Buenos Aires as the reference IRB. Recruiter Investigators The Recruiting Investigators must be gastroenterologists attending an adult population with a gastroenterology outpatient clinic that assists H. pylori infected patients. Before acceptance the outpatient clinic must attend, in a clinical routine basis, patients in which H. pylori diagnosis or treatment is indicated. Eradication confirmation tests have to be performed routinely. They will register the study variables of their own routine clinical practice in an e-CRF.

Study Variables Anonymised Patient Identifiers

Province/Centre/Investigator Gender Date of Birth Ethnic Background History and Comorbidity BMI Drug allergies Relevant comorbidities Current concomitant medication Data on Infection Indication for diagnosis and treatment Upper Gastrointestinal tract symptoms Diagnostic Test for current treatment Number and type of previous eradication attempts Prescribed Treatment Drugs Dosage and intakes per day Length of treatment Compliance Adherence to treatment (yes/no >90%) Probiotics use Adverse Events Type of event, intensity, duration and relation with treatment Treatment withdrawal due to adverse events. Efficacy Eradication (yes/no), test used, and date

ELIGIBILITY:
Inclusion Criteria:

Infected adult patients by Helicobacter pylori

-

Exclusion Criteria:

Pregnant or lactating women Subjects currently taking any antibiotics Administration of antibiotics or bismuth in the preceding 4 weeks or PPI 2 weeks previous Unable or refuse to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Infected adult patients by Helicobacter pylori
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2034-01-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of H pylori eradication regimens in the real world | At least 4-6 weeks after the treatment
  Eradication (yes or No). Negative Urea Breath Test or stool antigen

SECONDARY OUTCOMES:
Diagnostic methods for H pylori detection and eradication | 90 days
  Test used
Frecuency of adverse events | 90 days
  Any possible adverse events during the treatment period. Treatment withdrawal due to adverse events
Effectiveness of the different H pylori treatments according to BMI | 90 days
  BMI
Compliance rate | 90 days
  Compliance was defined as good when subjects had taken more than 90% of the total medication

CONTACTS AND LOCATIONS:
Overall Officials: Oscar M Laudanno, MD, Study Chair — Instituto de Investigaciones Médicas Alfredo Lanari. Universidad de Buenos Aires
Locations (1):
- Instituto de Investigaciones Medicas Alfredo Lanari. Universidad de Buenos Aires, Ciudad de Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share information during Digestive Congress and to publicate the results
Time Frame: As soon as we have new data
Access Criteria: Undecided

REFERENCES:
- [Result] Laudanno O, Ahumaran G, Gollo P, Khoury M, Thome M, Gonzalez P. Tailored Helicobacter pylori eradication therapy in obese patients undergoing bariatric surgery. Rev Esp Enferm Dig. 2021 May;113(5):345-347. doi: 10.17235/reed.2020.7433/2020. PMID 33244981
- See also: Instituto de Investigaciones Médicas Alfredo Lanari. University of Buenos Aires — http://lanari.uba.ar